CLINICAL TRIAL: NCT02425163
Title: Shear Wave Elastography of Prostate Cancer
Acronym: ElaProC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Johann J. Wendler, MD, Dr. med., University of Magdeburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD-URO-0047
Record Dates: First submitted 2015-02-10; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Shear Wave Elastography; Prostate; Prostate Biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- suspicious for Prostate Cancer (Active Comparator): PSA >4ng/ml or PSA-Velocity >0.75ng/ml/a or suspicious rectal examination or Status after external beam therapy of the prostate in prostate cancer.
  Patients who are able for transrectal ultrasound examination. Transrectal shear wave elastography of the prostate for Transrectal random biopsy of the prostate.
  Interventions: Device: Transrectal shear wave elastography of the prostate; Procedure: Transrectal random biopsy of the prostate

INTERVENTIONS:
Device: Transrectal shear wave elastography of the prostate — Transrectal shear wave elastography of the prostate with SuperSonic Imagine Ultrasound System AIXPLORER and an endocavity sonic head SE12-3 (SuperSonic Imagine, Aix-en-Provence, France)
  Other Names: SuperSonic Imagine Ultrasound System
Procedure: Transrectal random biopsy of the prostate — TRUS-SWE-guided random biopsies of the Prostata with 18G-gun
  Other Names: TRUS-SWE-guided random biopsies of the prostata

SUMMARY:
Evaluation of significant Shear Wave Elastography Parameters for Prostate Biopsy and Prostate Cancer detection.

DETAILED DESCRIPTION:
This Study will evaluate the Shear Wave Elastography (SWE) Parameters for Prostate Biopsy and Prostate Cancer detection.

ELIGIBILITY:
Inclusion Criteria:

* Suspicious for prostate cancer with no pretreatment and Prostata specific Antigen (PSA) >4ng/ml or PSA velocity > 0.75 ng/ml per year or suspicious transrectal digital examination
* Status after external beam radiotherapy of the prostate in localized prostate cancer and suspicious for local prostate cancer recurrence

Exclusion Criteria:

* None.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Shear wave elastography | 12 Months
  transrectal shear wave elastography with detection of prostate tissue pressure [kilo-Pascal] in correspondence to biopsy areas

SECONDARY OUTCOMES:
Differentiation of Entity by Elastography | 12 Months
  Elasticity and location of benign (normal, benign prostate hyperplasia) or malignant tissue (Prostate Cancer)
Differentiation of benign tissue elasticity depending on prostate Location (Basis, Mid, Apex) | 12 Months
  Differentiation of benign tissue elasticity depending on prostate Location (Basis, Mid, Apex)
Differentiation of Prostate cancer malignity by Elastography | 12 Months
  Differentiation of low-risk versus intermediate and high-risk Prostate cancer malignity (Gleason score 6 vs. 7-10) by Elastography
Histopathological Analysis | 12 Months
  Histopathological Analysis of biopsy specimen: benign prostate hyperplasia

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schostak, Prof. Dr., Principal Investigator — Urologische Klinik, Otto-von-Guericke University Magdeburg
Locations (1):
- Department of Urology University Hospital Otto-von-Guericke-University Magdeburg, Magdeburg, Saxony-Anhalt, Germany

REFERENCES:
- [Result] Correas JM, Tissier AM, Khairoune A, Vassiliu V, Mejean A, Helenon O, Memo R, Barr RG. Prostate cancer: diagnostic performance of real-time shear-wave elastography. Radiology. 2015 Apr;275(1):280-9. doi: 10.1148/radiol.14140567. Epub 2014 Nov 19. PMID 25599156